CLINICAL TRIAL: NCT03074318
Title: A Phase I/II Trial Combining Avelumab and Trabectedin for Advanced Liposarcoma and Leiomyosarcoma
Brief Title: Avelumab and Trabectedin in Treating Patients With Liposarcoma or Leiomyosarcoma That is Metastatic or Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to PI leaving institution
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); EMD Serono (Industry)
Responsible Party: Principal Investigator, Seth Pollack, Associate Professor of Medicine (Hematology and Oncology), Northwestern University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 9717; NCI-2017-00234 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9717 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG9217009 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-03-01; First posted 2017-03-08 (Actual); Results first posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Leiomyosarcoma; Metastatic Liposarcoma; Unresectable Leiomyosarcoma; Unresectable Liposarcoma
MeSH Terms: conditions — Leiomyosarcoma; Liposarcoma | interventions — avelumab; Trabectedin

STUDY DESIGN:
Intervention Model Description: Subjects were enrolled into Phase 1, first into 1.5 mg/m^2 trabectedin dose, then 1.0 mg/m^2 trabectedin, then 1.2 mg/m^2 trabectedin. Once the recommended Phase 2 dose was selected at 1.0 mg/m^2 trabectedin, all subsequent subjects were enrolled into Phase 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 (1.5 mg/m^2 trabectedin + avelumab) (Experimental): Avelumab will be administered every 2 weeks. Trabectedin will be administered every 3 weeks for the first two doses (Week 1 and Week 4), and then every four weeks (Week 7, Week 11,…) moving forward. After Cycle 2 of trabectedin, dosing may extend to every 5 weeks at investigator discretion, for management of trabectedin-associated toxicity only. Delays of trabectedin beyond 5 weeks may be allowed but require written approval from the Sponsor-Investigator. On days where both drugs are scheduled to be administered, avelumab will be administered first. This will continue until unacceptable toxicity or confirmed disease progression.
  Interventions: Drug: Avelumab; Drug: Trabectedin
- Phase 1 (1.0 mg/m^2 trabectedin + avelumab) (Experimental): Avelumab will be administered every 2 weeks. Trabectedin will be administered every 3 weeks for the first two doses (Week 1 and Week 4), and then every four weeks (Week 7, Week 11,…) moving forward. After Cycle 2 of trabectedin, dosing may extend to every 5 weeks at investigator discretion, for management of trabectedin-associated toxicity only. Delays of trabectedin beyond 5 weeks may be allowed but require written approval from the Sponsor-Investigator. On days where both drugs are scheduled to be administered, avelumab will be administered first. This will continue until unacceptable toxicity or confirmed disease progression.
  Interventions: Drug: Avelumab; Drug: Trabectedin
- Phase 1 (1.2 mg/m^2 trabectedin + avelumab) (Experimental): Avelumab will be administered every 2 weeks. Trabectedin will be administered every 3 weeks for the first two doses (Week 1 and Week 4), and then every four weeks (Week 7, Week 11,…) moving forward. After Cycle 2 of trabectedin, dosing may extend to every 5 weeks at investigator discretion, for management of trabectedin-associated toxicity only. Delays of trabectedin beyond 5 weeks may be allowed but require written approval from the Sponsor-Investigator. On days where both drugs are scheduled to be administered, avelumab will be administered first. This will continue until unacceptable toxicity or confirmed disease progression.
  Interventions: Drug: Avelumab; Drug: Trabectedin
- Phase 2 (1.0 mg/m^2 trabectedin + avelumab) (Experimental): Avelumab will be administered every 2 weeks. Trabectedin will be administered every 3 weeks for the first two doses (Week 1 and Week 4), and then every four weeks (Week 7, Week 11,…) moving forward. After Cycle 2 of trabectedin, dosing may extend to every 5 weeks at investigator discretion, for management of trabectedin-associated toxicity only. Delays of trabectedin beyond 5 weeks may be allowed but require written approval from the Sponsor-Investigator. On days where both drugs are scheduled to be administered, avelumab will be administered first. This will continue until unacceptable toxicity or confirmed disease progression.
  Interventions: Drug: Avelumab; Drug: Trabectedin

INTERVENTIONS:
Drug: Avelumab — Given IV
  Other Names: Bavencio; MSB-0010718C; MSB0010718C
Drug: Trabectedin — Given IV
  Other Names: Ecteinascidin; ecteinascidin 743; ET-743; Yondelis

SUMMARY:
This phase I/II studies the side effects of avelumab and trabectedin and how well they work in treating patients with leiomyosarcoma or liposarcoma that has spread to other places in the body (metastatic) or cannot be removed by surgery. Immunotherapy with monoclonal antibodies, such as avelumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as trabectedin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving avelumab and trabectedin may work better in treating patients with liposarcoma or leiomyosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of the combination of trabectedin and avelumab in subjects with advanced leiomyosarcoma and liposarcoma.

II. To assess the objective response rate of advanced L-type sarcoma patients receiving the combination regimen of avelumab and trabectedin.

SECONDARY OBJECTIVE:

I. To further explore the clinical activity and safety profile of avelumab and trabectedin as a combination therapy.

OUTLINE:

Avelumab will be administered every 2 weeks. Trabectedin will be administered every 3 weeks for the first two doses (Week 1 and Week 4), and then every four weeks (Week 7, Week 11,…) moving forward. After Cycle 2 of trabectedin, dosing may extend to every 5 weeks at investigator discretion, for management of trabectedin-associated toxicity only. Delays of trabectedin beyond 5 weeks may be allowed but require written approval from the Sponsor-Investigator. On days where both drugs are scheduled to be administered, avelumab will be administered first. This will continue until unacceptable toxicity or confirmed disease progression.

After completion of study treatment, patients are followed up at 30 and 90 days, then every 12 weeks for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Must have a histologically confirmed diagnosis of advanced (metastatic or unresectable) soft tissue sarcoma with one of the following subtypes:

  * Leiomyosarcoma
  * Liposarcoma
* Subject must be clinically indicated to receive trabectedin therapy as part of routine care. Subjects may be first line, or have received any number of prior systemic therapies
* Total bilirubin level =< 1.5 x the upper limit of normal (ULN) mg/dL
* Aspartate aminotransferase (AST) =< 2.5 x ULN and alanine aminotransferase (ALT) =< 2.5 x ULN
* Alkaline phosphatase < 2.5 x ULN
* Serum creatinine =< 1.5 x ULN
* Calculated creatinine clearance >= 30 mL/min using the Cockcroft-Gault formula may be included
* Creatinine phosphokinase (CPK) =< 2.5 x ULN
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelet count >= 100,000/mm^3 (100 x 10^9/L)
* Hemoglobin >= 9 g/dL
* Subject must demonstrate a left ventricular ejection fraction (LVEF) > 45% by echocardiography (ECHO) or multigated acquisition scan (MUGA)
* Male or non-pregnant and non-breast feeding female:

  * Females of child-bearing potential must agree to use highly effective contraception without interruption from initiation of therapy and while on study medication and have a negative serum pregnancy test (beta - human chorionic gonadotropin [hCG]) result at screening and agree to ongoing pregnancy testing during the course of the study, and at the end of study treatment; a highly effective method of contraception is defined as one that results in a low failure rate (that is, < 1% per year), when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, or a vasectomized partner
  * Male subjects must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study
* All ongoing toxicities related to prior therapies must be resolved to grade 1 or better (except alopecia)
* Subject must have an Eastern Cooperative Oncology Group (ECOG) performance status =< 1 or Karnofsky performance scale >= 70
* Subjects must have one or more measurable lesions, as determined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 assessed by computed tomography (CT) or magnetic resonance imaging (MRI)
* Subjects must have a life expectancy of >= 6 months, as determined by the treating physician
* Ability to understand and sign informed consent document
* Willingness and ability to comply with the scheduled visits, laboratory tests, and other study procedures

Exclusion Criteria:

* Known active, uncontrolled, or symptomatic central nervous system (CNS) metastases; a subject with controlled and asymptomatic CNS metastases may participate in this study; as such, the subject must have completed any prior treatment for CNS metastases >= 28 days (including radiotherapy and/or surgery) prior to the start of treatment in this study and should not be receiving chronic corticosteroid therapy in excess of 10 mg daily prednisone (or equivalent) for CNS metastases; subjects with known CNS metastases must be confirmed radiographically stable by at least one imaging study, at least 28 days from last treatment
* Receipt of any type of cytotoxic, biologic, or other systemic anticancer therapy (including investigational) within 2 weeks of enrollment
* Prior organ transplantation, including allogeneic stem cell transplantation
* Prior treatment with trabectedin
* Significant acute or chronic infections including, among others:

  * Known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
  * Known active infection with hepatitis B or hepatitis C
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:

  * Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
  * Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses =< 10 mg or 10 mg equivalent prednisone per day
  * Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, introocular, or inhalation) are acceptable
* Known severe hypersensitivity reactions to monoclonal antibodies (grade >= 3 National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5.0), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
* Pregnant or lactating females
* Known, active alcohol or drug abuse
* All other significant diseases (for example, inflammatory bowel disease, uncontrolled asthma), which, in the opinion of the investigator, might impair the subject's tolerance of trial treatment
* Any vaccination within 4 weeks of the first dose of avelumab, with the following exceptions:

  * Administration of inactivated vaccines, including inactivated flu vaccines, are allowable; however, they should not be given within 2 weeks prior to starting study treatment
* Clinically significant cardiovascular disease including cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), congestive heart failure with New York Heart Association (NYHA) class II or greater or serious cardiac arrhythmia requiring medication
* Severe (requiring active treatment) acute or chronic medical conditions including: colitis, inflammatory bowel disease, pneumonitis, or pulmonary fibrosis
* Recent (within the past year) or active suicidal ideation or behavior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Pollack, Principal Investigator — Northwestern University
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose Level 1: Subjects received 1.5 mg/m^2 of trabectedin plus avelumab.
- Phase 1 Dose Level 2: Subjects received 1.0 mg/m^2 of trabectedin plus avelumab
- Phase 1 Dose Level 3: Subjects received 1.2 mg/m^2 of trabectedin plus avelumab.
- Phase 2: Subjects received 1.0 mg/m^2 trabectedin plus avelumab.
Period: Overall Study
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 2
Started | 6 | 7 | 6 | 16
Completed | 2 | 2 | 0 | 0
Not Completed | 4 | 5 | 6 | 16
Not completed — Adverse Event | 0 | 1 | 1 | 1
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 4
Not completed — Trial Closure | 2 | 2 | 3 | 11

BASELINE CHARACTERISTICS:
Groups:
- Phase 1 (1.5 mg/m^2 Trabectedin); Phase 1 (1.0 mg/m^2 Trabectedin); Phase 1 (1.2 mg/m^2 Trabectedin): Phase 1: Avelumab will be administered every 2 weeks. Trabectedin will be administered every 3 weeks for the first two doses (Week 1 and Week 4), and then every four weeks (Week 7, Week 11,…) moving forward. After Cycle 2 of trabectedin, dosing may extend to every 5 weeks at investigator discretion, for management of trabectedin-associated toxicity only. Delays of trabectedin beyond 5 weeks may be allowed but require written approval from the Sponsor-Investigator. On days where both drugs are scheduled to be administered, avelumab will be administered first. This will continue until unacceptable toxicity or confirmed disease progression.
  Avelumab: Given IV
  Trabectedin: Given IV
- Phase 2 (Avelumab, Trabectedin): Phase 2: Avelumab will be administered every 2 weeks. Trabectedin will be administered every 3 weeks for the first two doses (Week 1 and Week 4), and then every four weeks (Week 7, Week 11,…) moving forward. After Cycle 2 of trabectedin, dosing may extend to every 5 weeks at investigator discretion, for management of trabectedin-associated toxicity only. Delays of trabectedin beyond 5 weeks may be allowed but require written approval from the Sponsor-Investigator. On days where both drugs are scheduled to be administered, avelumab will be administered first. This will continue until unacceptable toxicity or confirmed disease progression.
  Avelumab: Given IV
  Trabectedin: Given IV
- Total: Total of all reporting groups
Arm/Group | Phase 1 (1.5 mg/m^2 Trabectedin) | Phase 1 (1.0 mg/m^2 Trabectedin) | Phase 1 (1.2 mg/m^2 Trabectedin) | Phase 2 (Avelumab, Trabectedin) | Total
Number analyzed (Participants) | 6 | 7 | 6 | 16 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 4 | 7 | 22
  >=65 years | 2 | 0 | 2 | 9 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 3 | 11 | 20
  Male | 5 | 2 | 3 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 7 | 6 | 14 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1 | 2
  Asian | 0 | 1 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 4 | 5 | 12 | 27
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Type of Sarcoma [Count of Participants; unit: Participants]
  Uterine Leiomyosarcoma | 0 | 3 | 0 | 3 | 6
  Non-Uterine Leiomyosarcoma | 4 | 2 | 2 | 10 | 18
  Dedifferentiated Liposarcoma | 2 | 1 | 3 | 3 | 9
  Myxoid/Round Cell Liposarcoma | 0 | 1 | 0 | 0 | 1
  Pleomorphic Liposarcoma | 0 | 0 | 1 | 0 | 1
Lines of Prior Therapy [Count of Participants; unit: Participants]
  0 Lines of Prior Therapy | 2 | 0 | 0 | 3 | 5
  1 Line of Prior Therapy | 1 | 1 | 2 | 8 | 12
  2 Lines of Prior Therapy | 2 | 0 | 2 | 3 | 7
  3 Lines of Prior Therapy | 1 | 1 | 2 | 1 | 5
  4 Lines of Prior Therapy | 0 | 4 | 0 | 0 | 4
  5 Lines of Prior Therapy | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Measured by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Time Frame: up to 2 years 7 months total
Population: Cumulative number of adverse events experienced on trial by all patients, reported per grade.
Measure: Number; unit: number of adverse events
Groups:
- Phase 1 - 1.5 mg/m^2 Trabectedin: Subjects received 1.5 mg/m2 of trabectedin plus avelumab.
- Phase 1 - 1.0 mg/m^2 Trabectedin; Phase 2 - 1.0 mg/m^2 Trabectedin: Subjects received 1.0 mg/m^2 trabectedin plus avelumab.
- Phase 1 - 1.2 mg/m^2 Trabectedin: Subjects received 1.2 mg/m^2 trabectedin plus avelumab.
Arm/Group | Phase 1 - 1.5 mg/m^2 Trabectedin | Phase 1 - 1.0 mg/m^2 Trabectedin | Phase 1 - 1.2 mg/m^2 Trabectedin | Phase 2 - 1.0 mg/m^2 Trabectedin
Number analyzed (Participants) | 6 | 7 | 6 | 16
number of adverse events
  Grade 1 | 95 | 98 | 86 | 201
  Grade 2 | 41 | 46 | 33 | 115
  Grade 3 | 12 | 14 | 9 | 40
  Grade 4 | 2 | 0 | 0 | 6
  Grade 5 | 1 | 0 | 0 | 0

2. Primary Outcome: Overall Response Rate (ORR)
Description: Rate of Partial Response (PR) + Complete Response (CR), which is the best response for each subject determined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 for target lesions and assessed by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) scan. Partial response is defined as a decrease in 30% or more in the sum of the longest diameter of target lesions, and complete response is defined as disappearance of all evaluable disease. No subjects had a complete response on this study so the ORR represents subjects who had a partial response only.
Time Frame: Up to 2 years 7 months total
Population: Subjects enrolled in Phase 2 plus subjects treated at the Recommended Phase 2 Dose (RP2D).
Measure: Number; unit: percentage of participants
Groups:
- Treatment (Avelumab, Trabectedin): Subjects enrolled in Phase 2 plus subjects treated at the Recommended Phase 2 dose.
Arm/Group | Treatment (Avelumab, Trabectedin)
Number analyzed (Participants) | 23
percentage of participants | 13

3. Secondary Outcome: Time to Response
Description: Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Time to response is defined as the amount of time from when the subject first received study treatment (Cycle 1, Day 1) to when they achieved a partial response on trial.
  With such small numbers, this data is not necessarily representative of what a larger study would report.
Time Frame: Up to 2 years 7 months total
Population: Average time to response for the 4 subjects who responded in both Phase 1 and Phase 2. Only subjects who had a response to treatment are included in this analysis.
Measure: Mean (Full Range); unit: days
Groups:
- Phase 1 - 1.5 mg/m^2 Trabectedin; Phase 1 - 1.0 mg/m^2 Trabectedin; Phase 1 - 1.2 mg/m^2 Trabectedin; Phase 2 - 1.0 mg/m^2 Trabectedin: Avelumab will be administered every 2 weeks. Trabectedin will be administered every 3 weeks for the first two doses (Week 1 and Week 4), and then every four weeks (Week 7, Week 11,…) moving forward. After Cycle 2 of trabectedin, dosing may extend to every 5 weeks at investigator discretion, for management of trabectedin-associated toxicity only. Delays of trabectedin beyond 5 weeks may be allowed but require written approval from the Sponsor-Investigator. On days where both drugs are scheduled to be administered, avelumab will be administered first. This will continue until unacceptable toxicity or confirmed disease progression.
  Avelumab: Given IV
  Trabectedin: Given IV
Arm/Group | Phase 1 - 1.5 mg/m^2 Trabectedin | Phase 1 - 1.0 mg/m^2 Trabectedin | Phase 1 - 1.2 mg/m^2 Trabectedin | Phase 2 - 1.0 mg/m^2 Trabectedin
Number analyzed (Participants) | 1 | 0 | 0 | 3
days | 158 |  |  | 189 [77 to 329]

4. Secondary Outcome: Duration of Response
Description: Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Duration of response is defined as the amount of time a subject responded to study treatment with either a partial response or complete response until the date of last follow-up (if response ongoing at data cutoff) or the date until they progressed on study.
Time Frame: Up to 2 years 7 months total
Population: Average duration of response for the 4 subjects who responded to treatment in both Phase 1 and Phase 2. Only subjects who had a response to treatment are included in this analysis.
Measure: Mean (Full Range); unit: days
Arm/Group | Phase 1 - 1.5 mg/m^2 Trabectedin | Phase 1 - 1.0 mg/m^2 Trabectedin | Phase 1 - 1.2 mg/m^2 Trabectedin | Phase 2 - 1.0 mg/m^2 Trabectedin
Number analyzed (Participants) | 1 | 0 | 0 | 3
days | NA — Data not representative of actual duration of response due to low response rate overall, late time to response for 1 subject, and study closing early while subjects still responding. |  |  | NA [NA to NA] — Data not representative of actual duration of response due to low response rate overall, late time to response for 1 subject, and study closing early while subjects still responding.

5. Secondary Outcome: Progression-free Survival (PFS)
Description: Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Progression is defined using RECIST v1.1, as a 20% increase in the sum of the longest diameter of target lesions, appearance of new lesions while on study, or clear growth of a non-target lesion.
Time Frame: At 12 weeks
Population: All subjects treated in Phase 1 and Phase 2 evaluated at 3 months. NOTE: one subject was not evaluable for response and was replaced after withdrawing from study before response evaluation.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 - 1.5 mg/m^2 Trabectedin | Phase 1 - 1.0 mg/m^2 Trabectedin | Phase 1 - 1.2 mg/m^2 Trabectedin | Phase 2 - 1.0 mg/m^2 Trabectedin
Number analyzed (Participants) | 6 | 6 | 6 | 16
percentage of participants | 50 | 50 | 83 | 63

6. Secondary Outcome: Complete Response Rate (CR)
Description: Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete Response is defined as disappearance of all evaluable disease.
Time Frame: At 12 weeks
Population: NOTE: one subject was not evaluable for response and was replaced after withdrawing from study before response evaluation.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1, 1.5 mg/m^2 Trabectedin; Phase 1, 1.0 mg/m^2 Trabectedin; Phase 1, 1.2 mg/m^2 Trabectedin; Phase 2, 1.0 mg/m^2 Trabectedin: Avelumab will be administered every 2 weeks. Trabectedin will be administered every 3 weeks for the first two doses (Week 1 and Week 4), and then every four weeks (Week 7, Week 11,…) moving forward. After Cycle 2 of trabectedin, dosing may extend to every 5 weeks at investigator discretion, for management of trabectedin-associated toxicity only. Delays of trabectedin beyond 5 weeks may be allowed but require written approval from the Sponsor-Investigator. On days where both drugs are scheduled to be administered, avelumab will be administered first. This will continue until unacceptable toxicity or confirmed disease progression.
  Avelumab: Given IV
  Trabectedin: Given IV
Arm/Group | Phase 1, 1.5 mg/m^2 Trabectedin | Phase 1, 1.0 mg/m^2 Trabectedin | Phase 1, 1.2 mg/m^2 Trabectedin | Phase 2, 1.0 mg/m^2 Trabectedin
Number analyzed (Participants) | 6 | 6 | 6 | 16
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Partial Response Rate (PR)
Description: Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Partial response is defined as a decrease in 30% or more in the sum of the longest diameter of target lesions.
Time Frame: At 12 weeks
Population: NOTE: One subject was not evaluable for response and was replaced after withdrawing from the study before response evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - 1.5 mg/m^2 Trabectedin | Phase 1 - 1.0 mg/m^2 Trabectedin | Phase 1 - 1.2 mg/m^2 Trabectedin | Phase 2 - 1.0 mg/m^2 Trabectedin
Number analyzed (Participants) | 6 | 6 | 6 | 16
Participants | 1 | 0 | 0 | 3

8. Secondary Outcome: Stable Disease (SD)
Description: Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Stable Disease is defined as neither sufficient shrinkage to qualify for a Partial Response (PR) nor sufficient increase to qualify for Progressive Disease (PD).
Time Frame: At 12 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - 1.5 mg/m^2 Trabectedin | Phase 1 - 1.0 mg/m^2 Trabectedin | Phase 1 - 1.2 mg/m^2 Trabectedin | Phase 2 - 1.0 mg/m^2 Trabectedin
Number analyzed (Participants) | 6 | 6 | 6 | 16
Participants | 2 | 3 | 4 | 7

9. Secondary Outcome: Clinical Benefit Rate
Description: Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Clinical Benefit Rate is defined as the percentage of subjects who achieved a Complete Response (CR) + Partial Response (PR) + Stable Disease (SD).
Time Frame: At 12 weeks
Population: Subjects with a Partial Response (PR) or Stable Disease (SD) treated at the RP2D. No subjects achieved a Complete Response (CR) while on study.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Avelumab, Trabectedin)
Number analyzed (Participants) | 23
percentage of participants | 56

10. Secondary Outcome: Median Overall Survival (OS)
Description: Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: Up to 2 years post End of Treatment, for a total of 3 years
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Phase 1 - 1.5 mg/m^2 Trabectedin | Phase 1 - 1.0 mg/m^2 Trabectedin | Phase 1 - 1.2 mg/m^2 Trabectedin | Phase 2 - 1.0 mg/m^2 Trabectedin
Number analyzed (Participants) | 6 | 7 | 6 | 16
days | 391 [22 to 759] | 416 [0 to 906] | NA [NA to NA] — The study was closed early when Principal Investigator left institution, so outcome was not reached for this cohort. | NA [NA to NA] — The study was closed early when Principal Investigator left institution, so outcome was not reached for this cohort.

11. Secondary Outcome: Adverse Event Profile - All Treatment-Related Grade 3-5 Adverse Events
Description: Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Time Frame: Up to 2 years 7 months total
Measure: Number; unit: Events
Arm/Group | Phase 1 - 1.5 mg/m^2 Trabectedin | Phase 1 - 1.0 mg/m^2 Trabectedin | Phase 1 - 1.2 mg/m^2 Trabectedin | Phase 2 - 1.0 mg/m^2 Trabectedin
Number analyzed (Participants) | 6 | 7 | 6 | 16
Events
  Alanine Aminotransferase Increased | 1 | 1 | 1 | 3
  Lymphocyte Count Decreased | 0 | 0 | 0 | 4
  Neutrophil Count Decreased | 1 | 2 | 0 | 0
  Anemia | 0 | 0 | 0 | 2
  Ejection Fraction Decreased | 1 | 0 | 1 | 0
  Aspartate Aminotransferase Increased | 0 | 0 | 0 | 1
  Blood Bilirubin Increased | 1 | 0 | 0 | 0
  Dyspnea | 0 | 0 | 0 | 1
  Fatigue | 0 | 0 | 0 | 1
  Gastrointestinal Disorders - Other | 0 | 1 | 0 | 0
  GGT Increased | 1 | 0 | 0 | 0
  Hepatobiliary Disorders - Other | 1 | 0 | 0 | 0
  Hypophosphatemia | 1 | 0 | 0 | 0
  Infections and Infestations - Other (Port Infection/Inflammation/Erythema) | 1 | 0 | 0 | 0
  Infusion Related Reaction | 0 | 0 | 0 | 1
  Muscle Weakness Lower Limb | 0 | 0 | 0 | 1
  Respiratory Failure | 1 | 0 | 0 | 0
  Syncope | 1 | 0 | 0 | 0
  White Blood Cell Decreased | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE) will be monitored from the time of first exposure to study drug (Cycle 1 Day 1) through 90 days following the last dose of a study drug, up to 2 years 7 months total. All-cause mortality was assessed from enrollment to end of study or subject death, up to 3 years total.
Groups:
- Phase 1 - 1.0 mg/m^2 Trabectedin; Phase 1 - 1.2mg/m^2 Trabectedin: Avelumab will be administered every 2 weeks. Trabectedin will be administered every 3 weeks for the first two doses (Week 1 and Week 4), and then every four weeks (Week 7, Week 11,…) moving forward. After Cycle 2 of trabectedin, dosing may extend to every 5 weeks at investigator discretion, for management of trabectedin-associated toxicity only. Delays of trabectedin beyond 5 weeks may be allowed but require written approval from the Sponsor-Investigator. On days where both drugs are scheduled to be administered, avelumab will be administered first. This will continue until unacceptable toxicity or confirmed disease progression.
Arm/Group | Phase 1 - 1.5 mg/m^2 Trabectedin | Phase 1 - 1.0 mg/m^2 Trabectedin | Phase 1 - 1.2mg/m^2 Trabectedin | Phase 2 - 1.0 mg/m^2 Trabectedin
All-Cause Mortality (participants affected / at risk) | 4/6 | 5/7 | 2/6 | 1/16
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/7 | 1/6 | 7/16
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 6/6 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 - 1.5 mg/m^2 Trabectedin (N=6) | Phase 1 - 1.0 mg/m^2 Trabectedin (N=7) | Phase 1 - 1.2mg/m^2 Trabectedin (N=6) | Phase 2 - 1.0 mg/m^2 Trabectedin (N=16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tricuspid valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Small intestinal obstruction
Gastrointestinal disorders - other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Acute Diverticulitis
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tricuspid valve mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LFT Elevation (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Hematemesis
Gastrointestinal disorders - other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Melena
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 - 1.5 mg/m^2 Trabectedin (N=6) | Phase 1 - 1.0 mg/m^2 Trabectedin (N=7) | Phase 1 - 1.2mg/m^2 Trabectedin (N=6) | Phase 2 - 1.0 mg/m^2 Trabectedin (N=16)
Fatigue (General disorders) | 6 (8) | 6 (6) | 5 (6) | 16 (19)
Nausea (Gastrointestinal disorders) | 6 (8) | 5 (5) | 3 (3) | 13 (14)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 4 (10) | 4 (6) | 6 (7)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 5 (6) | 8 (8)
Vomiting (Gastrointestinal disorders) | 5 (7) | 2 (4) | 3 (4) | 8 (9)
Alanine aminotransferase increase (Investigations) | 3 (5) | 1 (2) | 5 (7) | 6 (19)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (6) | 5 (5)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (5) | 5 (5)
Headache (Nervous system disorders) | 2 (2) | 2 (3) | 3 (3) | 4 (7)
Pain (General disorders) | 4 (6) | 2 (4) | 0 (0) | 4 (4)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 4 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 2 (2) | 8 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 2 (3) | 5 (10)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 0 (0) | 1 (1) | 5 (9)
Dizziness (Nervous system disorders) | 3 (3) | 1 (2) | 2 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1) | 6 (11)
Flu like symptoms (General disorders) | 1 (1) | 3 (6) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 11 (20)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (4) | 4 (4)
Creatinine Increaed (Investigations) | 2 (3) | 1 (1) | 0 (0) | 3 (5)
Fever (General disorders) | 2 (3) | 2 (3) | 0 (0) | 3 (8)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (3) | 3 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (3)
Chills (General disorders) | 1 (2) | 2 (3) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Dry Skin (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Blurred Vision (Eye disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2)
Alkaline Phosphatase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (9)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Non-cardiac chest pain (General disorders) | 1 (2) | 2 (3) | 0 (0) | 1 (1)
Nervous System Disorders - Other (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Infections and infestations - Other (Infections and infestations) | 3 (3) | 3 (3) | 3 (3) | 4 (5) — Port complications
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (9) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 1 (6) | 2 (4)
Edema limbs (General disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (2) | 1 (3)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (4)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest Pain - Cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tricuspid Valve Disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Watering Eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CPK increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INR Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Active Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiculitis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left Total Hip Dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucinations (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye Disorders - Other (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GGT increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Soreness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Heartburn
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concentration impairment (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body Aches (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorders - other (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - other (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infective myositis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sebaceous Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocrine Disorders - Other (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgical and Medical Procedures - Other (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scalp Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Disorders - Other (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT03074318/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT03074318/ICF_001.pdf